CLINICAL TRIAL: NCT01168778
Title: Improving Communication During Pediatric Visits for Acute Respiratory Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Rita Mangione-Smith, University of Washington/ Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 32542-A; 61-5957 (Other: Children's IRB application number)
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Upper Respiratory Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Behavioral: Physician Workshop

INTERVENTIONS:
Behavioral: Physician Workshop — Physicians that were assigned to the intervention group attended a 3.5 hour intervention workshop where they were trained in skills to communicate information about physical examination findings, treatment, and follow-up that will ultimately facilitate appropriate antibiotic prescribing and increase parent satisfaction with care.
  Arms: Intervention

SUMMARY:
The excessive use of outpatient antibiotics in the pediatric population has contributed to the rapid development of resistance in many strains of Streptococcus pneumoniae. Research has shown that community-based interventions may have a modest impact on reducing the injudicious use of antibiotics in children. However, since the actual prescribing of antibiotics is done by physicians and research has shown that physician-parent communication patterns during pediatric visits for acute respiratory tract infections (ARTI) strongly influence antibiotic prescription rate, it is crucial to develop effective interventions aimed specifically at them.

The overall goal of this study is to improve physician-parent communication patterns during visits for pediatric ARTI and, ultimately, to decrease rates of antibiotic prescribing for these illnesses in children.

DETAILED DESCRIPTION:
The overall goal of this study is to test a novel communication-based intervention aimed at decreasing rates of prescribing antibiotics for ARTI in children. We propose a randomized controlled trial involving a sample of 34 primary care pediatricians drawn from 8 practices in the Puget Sound Pediatric Research Network (PSPRN). Our research design incorporates a novel physician intervention that teaches the importance of specific physician communication behaviors. The primary physician outcomes for the study will be changes in the utilization of communication behaviors as reported by parents, and antibiotic prescribing rates for children presenting with ARTI symptoms. The primary parent outcome measure for the study will be satisfaction with care. Changes in the primary outcomes for the intervention physicians will be compared to changes in these outcomes for control physicians. The trial has five specific aims and five major hypotheses.

1. To evaluate the effectiveness of the proposed intervention in achieving its stated goals of changing physician communication behaviors.

   * We hypothesize that physicians in the intervention group will have increased reported use of desirable communication behaviors and decreased reported use of undesirable communication behaviors relative to control group physicians.
2. To determine the antibiotic prescribing rates for children aged 6 months to 10 years presenting with ARTI symptoms and assess how these rates change as a function of the intervention.

   * We hypothesize that physicians in the intervention group will decrease antibiotic prescribing rates for ARTI relative to the control group physicians.
3. To determine visit-specific satisfaction levels for parents of children seen by study physicians and assess how satisfaction levels change as a function of the intervention.

   * We hypothesize that parents who take their children to physicians in the intervention group will report increased satisfaction with care, relative to control group physicians.
4. To identify the factors (e.g., physician communication behaviors) that mediate the relationships between physicians being in the intervention group, decreased antibiotic prescribing, and increased parent satisfaction with care.

   * We hypothesize that increased use of desirable communication behaviors and decreased use of undesirable communication behaviors will partially mediate the relationships between being an intervention group physician, decreased inappropriate prescribing, and increased parent satisfaction with care.
5. To perform a validation study of the Physician Communication Behavior Inventory (PCBI) survey items. Using a standardized approach, specific physician communication behaviors will be coded through review of 100 video taped physician-parent encounters. The behaviors coded will be compared to parent responses on the PCBI surveys from these encounters.

   * We hypothesize that parent reports of physician communication behaviors on the PCBI will be highly correlated with actual physician communication behaviors coded from video tape data.

ELIGIBILITY:
Inclusion Criteria:

* Parents: the parent must present with a child between the ages of 6 months and 10 years old, who has not received antibiotics for any reason in the prior two weeks and who has any of the following symptoms: cough, runny nose/congestion, sore throat, ear pain, or ear tugging. Parents must be able to read English or Spanish; the visit must occur during one of the three data collection periods for the participating physician; and parents must have not previously participated in teh study.
* Physicians: physician must be a member of Puget Sound Pediatric research Network (PSPRN).

Exclusion Criteria:

* Parents: parents who are 18 years of age or less
* Physicians: physicians who are not members of PSPRN

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1313 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness of intervention in changing physician communication behaviors | 12 months
  To evaluate the effectiveness of the proposed intervention in achieving its stated goals of changing physician communication behavoirs

SECONDARY OUTCOMES:
Antibiotic prescribing rates as a function of the intervention | 12 months
  To determine the antibiotic prescribing rates for children aged 6 months to 10 years presenting with ARTI symptoms and assess how these rates change as a function of the intervention
Satisfaction levels for parents as a function of the intervention | 12 months
  To determine visit-specific satisfaction levels for parents of children seen by study physicians and assess how satisfaction levels change as a function of the intervention
Factor identification | 12 months
  To identify the factors (e.g., physician communication behaviors) that mediate the relationships between physicians being in the intervention group, decreased antibiotic prescribing, and increased parent satisfaction with care
Validation study of the PCBI | 12 months
  To perform a validation study of the Physician Communication Behavior Inventory (PCBI) survey items. Using a standardized approach, specific physician communication behaviors will be coded through review of 100 video taped physician-parent encounters. The behaviors coded will be compared to parent responses on the PCBI surveys from these encounters.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mangione-Smith, MD, MPH, Principal Investigator — University of Washington/ Seattle Children's Hospital; James A Taylor, MD, MPH, Principal Investigator — University of Washington